CLINICAL TRIAL: NCT00521859
Title: Dose Escalation Trial of Cloretazine (VNP40101M) and Hematopoietic Cell Transplantation for Patients With Selected, Poor-Prognosis Hematologic Malignancies
Brief Title: Cloretazine (VNP40101M) With Hematopoietic Cell Transplantation for Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Vion Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0844
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Hematologic Malignancies
Keywords: Hematologic Malignancies; Leukemia; Lymphoma; Myeloma; Hodgkin's Disease; Hematopoietic Cell Transplantation; Cloretazine; VNP40101M; Fludarabine; Fludarabine Phosphate; Fludara; ATG; Antithymocyte; Thymoglobulin
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Hodgkin Disease | interventions — laromustine; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cloretazine + Fludarabine (Experimental)
  Interventions: Drug: Cloretazine; Drug: Fludarabine

INTERVENTIONS:
Drug: Cloretazine — 800 mg/m^2 by vein daily
  Other Names: VNP40101M
Drug: Fludarabine — 25 mg/m^2 by vein daily x 5 Days
  Other Names: Fludarabine Phosphate; Fludara

SUMMARY:
Primary:

Define the maximal tolerated dose (MTD) of VNP40401M when given with hematopoietic cell transplantation (HCT)

Secondary:

* Describe the change in pharmacokinetic (PK) parameters with increasing doses of drug.
* Describe and estimate the frequency of > Grade 3 non-hematologic/non-infectious toxicities at the MTD.
* Report the efficacy of the regimen.
* Evaluate the rate of engraftment for the regimen.

DETAILED DESCRIPTION:
An autologous transplant uses the recipient's own stem cells, from the blood and bone marrow, for infusion.

VNP40101M is a chemotherapy drug designed to interfere with the growth and development of cancer cells, by binding to structures within cancer cells. This drug, given in higher doses, causes lowering of blood cells. Chemotherapy is commonly given to patients before a stem cell transplantation to help kill more cancer cells. After receiving this drug, stem cells are transfused (given gradually) to allow re-growth of the blood cells.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have blood drawn (about 3 tablespoons) for routine tests. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate). You will have a bone marrow biopsy. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of marrow and bone is withdrawn through a large needle. You will have a chest x-ray and computed tomography (CT) and positron emission tomography (PET) scans, if required, to measure your tumor. You will have a lung function test and an electrocardiogram (ECG-a test to measure the electrical activity of the heart). Women who are able to have children must have a negative blood or urine pregnancy test. If you will have a blood pregnancy test it will be done with routine blood tests.

Before you receive treatment on this study, you will have apheresis done to collect some of your stem cells. Apheresis is the process of removing part of the blood (such as platelets or white blood cells) from the body in order to remove certain elements, such as stem cells. Then the rest of the blood is returned back to the body. Your stem cells will be put back in your body after you finish treatment with VNP40101M. Apheresis will be done by a major vein through a central venous catheter (CVC), usually in the chest. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. The details of apheresis as well as the CVC will be described in separate consent forms. Your doctor will explain these procedures to you in more detail, and you will be required to sign a separate consent form for each procedure.

If you are found to be eligible to take part in this study, you will receive a dose of VNP40101M. The dose you receive will depend on when you enrolled in this study. The dose that you receive will remain the same throughout this study. Researchers will continue to enroll patients at the next highest dose level until the highest tolerable dose is found.

About 1 week after your stem cells are collected, you will be admitted to the hospital. You will stay in the hospital for about 3 weeks. You will then receive VNP40101M by a CVC over 6 hours.

Two days after you receive VNP40101M, the autologous stem cells (blood or bone marrow) will then be given to you by your CVC. You will receive G-CSF as an injection just under your skin daily, starting 1 week after your transplantation, which will help your blood cell levels return to normal.

You will then have blood drawn (about 5 tablespoons) for PK testing to measure the levels of VNP40101M in your blood. These samples will be drawn through a heparin lock, which will be in place for 24 hours after the study treatment is complete. A heparin lock is a small tube connected to a CVC in a vein in the arm for easy access. The heparin lock will be removed after these samples are received.

After you are released from the hospital, you will be required to stay in the Houston area for up to 1 month after the transplantation or until you are no longer experiencing any intolerable side effects. You will be asked to return to M. D. Anderson between 2-4 months following transplantation so that any late side effects of the study drug can be observed.

As part of standard care, you will have blood tests (about 3 tablespoons) for routine tests. Your health status will be followed-up to continue to check on the status of the disease. You will have a computed tomography scan and PET scan. You will also have a bone marrow biopsy.

If the disease gets worse or you experience any intolerable side effects, you will be taken off this study.

THIS IS AN INVESTIGATIONAL STUDY. VNP40101M is not FDA approved or commercially available. It is authorized for use in research only.

Up to 42 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years for autotransplant patients and age 18 to 60 years for allotransplant patients.
2. Patients with acute leukemia/MDS or lymphoid malignancies, including Hodgkin's and non-Hodgkin's lymphoma (primary refractory or refractory relapse), or multiple myeloma (beyond first remission or unresponsive to therapy), not qualifying for treatment protocols of higher priority.
3. Adequate renal function, as defined by serum creatinine <1.5 mg/dL.
4. Adequate hepatic function, as defined by SGPT <3 X upper limit of normal; serum bilirubin and alkaline phosphatase <2 X upper limit of normal, or considered not attributable to liver disease in the case of alkaline phosphatase.
5. Adequate pulmonary function with FEV1, FVC and DLCO >50% of expected corrected for hemoglobin.
6. Adequate cardiac function with left ventricular ejection fraction >40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
7. Zubrod performance status <2
8. Patients receiving an allogeneic transplant must have a related or unrelated donor which meets departmental standards for donor selection.

Exclusion Criteria:

1. Uncontrolled life-threatening infections
2. HIV positive
3. A positive Beta HCG in a woman with child bearing potential as defined as not being post-menopausal for 12 or more months or no previous surgical sterilization procedures.
4. Any CNS involvement which has not been controlled for at least 4 weeks
5. Patients must be at least 21 days from prior systemic therapy for their malignancy, or have improvement of all reversible toxicities to </= grade 2, whichever occurs first.
6. Any patient receiving Antabuse
7. Patients should be off metronidazole (Flagyl) for at least 24 hours prior to starting VNP40401M

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To study the highest tolerable dose of VNP40101M that can be given to patients with a form of leukemia, MDS, lymphoma, or myeloma in preparation for an autologous stem cell transplant. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Roy B. Jones, MD, PhD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org